CLINICAL TRIAL: NCT02089009
Title: Comparison of Non-mydriatic Camera Systems for Screening and Follow-up Examinations -Focused on the Retinal Vessel Situation- in the Population of a Female Health Hospital
Brief Title: Comparison of Non-mydriatic Camera Systems in a Female Health Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Martin Leitritz (Other)
Collaborators: Optomed (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Martin Leitritz, Dr. med. Martin A. Leitritz, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NonMydGyn
Record Dates: First submitted 2014-03-11; First posted 2014-03-17 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Eye Diseases; Retina; Lesion; Optic Disc Structural Anomaly
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Standard Population (Other): Retinal Imaging, vessel measurements, vessel changes of a population of a female health hospital
  Interventions: Other: Retinal imaging; Other: Vessel measurements; Other: Change in vessel diameters
- Group 2 Pregnant Population (Other): Change in vessel diameter at perinatal visits with retinal imaging (Retinal Imaging, vessel measurements, vessel changes)
  Interventions: Other: Retinal imaging; Other: Vessel measurements; Other: Change in vessel diameters

INTERVENTIONS:
Other: Retinal imaging — Retinal imaging by using non-mydriatic camera devices
Other: Vessel measurements — Vessel measurements based on the taken images by the use of a specialized software
Other: Change in vessel diameters — Change of vessel diameters before and after delivery based on the taken images by the use of a specialized software

SUMMARY:
1. To compare quality and usability of images taken by two different camera-systems without dilating the pupil.
2. To compare the retinal vessel diameters based on the images of to different camera-systems.
3. To detect changes in retinal vessel diameters while pregnancy and after delivery.

DETAILED DESCRIPTION:
1. To compare quality and usability of images taken by two different camera-systems without dilating the pupil.

   Quality means in this content that images cover the planned region of interest and images should be sharp and good illuminated to see details for medical reading of retinal findings.
2. To compare the retinal vessel diameters based on the images of to different camera-systems.

   The diameters of arteries and veins are planned to be measured with an automated software algorithm. Are there differences in the calculated results between the two used camera devices?
3. To detect changes in retinal vessel diameters while pregnancy and after delivery.

Are there detectable changes of the retinal findings between the images taken before and after delivery (e.g. bleeding, edema, vessel tortuosity)

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age >18 years
* pregnancy (only group 2)

Exclusion Criteria:

* limited ability for agreement
* heavy tremble
* reduced general condition
* known epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Image Quality | 12 to 16 month
  Visit 1 and Visit 2 (for group 2) Evaluating of image quality for each camera-system

SECONDARY OUTCOMES:
Retinal Pathologies | 12 to 16 month
  Visit 1 and Visit 2 (group 2) Which pathologies / diseases can be assessed with the taken images.
Differences Perinatal | 12 to 16 month
  Visit 1 and Visit 2 (group 2)

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Leitritz, M.D., Principal Investigator — University Hospital Tuebingen
Locations (2):
- Germany (2):
  - Female Health Hospital Reutlingen, Reutlingen, Baden-Wurttemberg
  - University Eye Hospital, Tübingen, Baden-Wurttemberg